CLINICAL TRIAL: NCT05064085
Title: A Phase I Trial of Capecitabine in Combination With Cemiplimab in Patients With Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Capecitabine In Combination With Cemiplimab In Patient With Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20902; R2810-ONC-20109 (Other: Regeneron Pharmaceuticals, Inc.)
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hormone Receptor-positive Breast Cancer
Keywords: Breast Cancer; HR+
MeSH Terms: conditions — Breast Neoplasms | interventions — cemiplimab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Level 1 (Experimental): Cemiplimab 350mg + Capecitabine 800 mg/m^2
  Interventions: Drug: Cemiplimab; Drug: Capecitabine
- Dose Level 2 (Experimental): Cemiplimab 350mg + Capecitabine 1000 mg/m^2
  Interventions: Drug: Cemiplimab; Drug: Capecitabine

INTERVENTIONS:
Drug: Cemiplimab — Participants will be given Cemiplimab 350 mg IV day 1 every 21 days
  Other Names: Libtayo
Drug: Capecitabine — Participants will take Capecitabine at 2 dose levels: 800 mg/m^2 and 1000 mg/m^2 by mouth twice daily 14 days on, 7 days off starting on day 3 every 21 days.
  Other Names: Xeloda

SUMMARY:
This is a single-center, open-label, phase I study to assess the safety and efficacy of the oral chemotherapy capecitabine in combination with cemiplimab in patients with hormone-receptor-positive (HR+) metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide a written informed consent and any locally required authorization prior to performing any protocol-related procedures,including screening evaluations.
* Female or male, age 18 years or older
* Eastern Cooperative Oncology Group (EGOG) performance status 0 through 2
* Pathologic confirmation of noninvasive breast cancer that is Hormone-receptor positive (HR+) (ER [estrogen-receptor] and/or PR [progesterone-receptor] >/= 1%, locally advanced, or metastatic disease.
* Invasive breast cancer is Human Epidermal Growth Factor Receptor 2 (HER2) negative defined as 0 or 1+ by immunohistochemistry (IHC) or with an in situ hybridization (ISH) ratio (HER2 gene copy/chromosome 17) < 2 or as defined by ASCO/CAP guidelines
* Measurable or non-measurable disease
* Any line of prior endocrine therapy in the unresectable and /or metastatic setting
* Adequate organ and marrow function as defined in protocol
* Participants must be willing and able to comply with the protocol for the duration of the study. This compliance includes undergoing treatment, scheduled visits, and examinations, including follow-up.
* If taking herbal or natural remedies that may have immune modulatory effects, participants must be willing to discontinue them before first dose of cemiplimab
* Body weight greater than 30 kg

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Received prior systemic cytotoxic chemotherapy for unresectable and/or metastatic disease. Patients who received 1 cycle or fewer at least 3 months prior to enrollment, which was discontinued for reasons other than disease progression, may be enrolled at the discretion of the PI.
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including cemiplimab.
* Nontreated brain metastasis. Treated brain metastasis is allowed if patients are stable and off steroids for at least 2 months prior to enrollment.
* Leptomeningeal disease.
* History of another primary malignancy, except for malignancy treated with curative intent; no known active disease for ≥2 years; adequately treated non-melanoma skin cancer or lentigo maligna (without evidence of disease); or adequately treated carcinoma in situ without evidence of disease (eg, cervical cancer in situ).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of cemiplimab, with the exceptions of intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection); systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid; or steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, pneumonitis etc]). The following are exceptions to this criterion: (a) Patients with vitiligo or alopecia. (b) Patients with hypothyroidism (eg, following Hashimoto syndrome) who are stable on hormone replacement. (c) Any chronic skin condition that does not require systemic therapy. (d) Patients without active disease in the last 5 years may be included but only after consultation with the study physician. (e) Patients with celiac disease controlled by diet alone.
* Prior treatment with other immune-modulating agents that was (a) within fewer than 4 weeks (28 days) prior to the first dose of cemiplimab or (b) associated with immune-mediated AEs that were ≥ grade 1 within 90 days prior to the first dose of cemiplimab or (c) associated with toxicity that resulted in discontinuation of the immune-modulating agent
* Prior treatment with idelalisib. The decision to treat with cemiplimab tumor types for which cemiplimab and/or other anti-PD-1/ PD-L1 agents have demonstrated efficacy, such as advanced CSCC, merits an individualized risk:benefit assessment by the treating physician in discussion with the patient, in the event that a patient had prior exposure to idelalisib.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* Known allergy or history of hypersensitivity to cemiplimab or any excipient.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for the hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Note: This is applied only to patients with a known infection. Screening tests for TB, hepatitis B and C, or HIV are not required.
* Receipt of live attenuated vaccination within 30 days prior to receiving cemiplimab. Note: Patients, if enrolled, should not receive a live vaccine while receiving cemiplimab and up to 30 days after the last dose of cemiplimab.
* Any condition that, in the opinion of the investigator, would interfere with the evaluation of the study treatment or interpretation of patient safety or study results.
* Patients with uncontrolled seizures.
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of investigational product.
* Patient is currently pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 24 months
  Recommended Phase 2 dose of Capecitabine combined with Cemiplimab will be determined by testing 2 dose levels. RP2D reflects the highest dose that did not cause Dose Limiting Toxicity (DLT)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  Objective response rate is defined as the sum of complete response and partial response based on Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1.
Clinical Benefit Rate (CBR) | Up to 24 months
  Clinical benefit rate is defined as the sum of complete response, partial response, and stable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1.
Progression Free Survival (PFS) | Up to 24 months
  Progression free survival is defined as the time from start of treatment to documented disease progression or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Aixa E Soyano Muller, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aixa Elena Soyano Muller et al. Phase I trial of capecitabine with cemiplimab in patients with hormone receptor-positive metastatic breast cancer.. JCO 43, e13082-e13082(2025). DOI:10.1200/JCO.2025.43.16_suppl.e13082